CLINICAL TRIAL: NCT04853810
Title: CUTADIAB OBSERVATORY Investigation of the Skin Manifestations Associated With the Adhesives of Technological Tools for Diabetes
Brief Title: Skin Manifestations Associated With Adhesives in Diabetes Technology Tools
Acronym: CUTADIAB
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200089; 2019-A03208-49 (Other: IDRCB)
Record Dates: First submitted 2021-02-26; First posted 2021-04-21 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major diabetic subjects having used a system with adhesives: Major diabetic subjects, whatever the etiology of diabetes, using or having used in the last 10 years a system with skin adhesives, i.e. insulin patch pump (e.g. OMNIPOD®, cell Novo®), pump with externalized catheter (e.g. MINIMED 640G®, YpsoPump®) or continuous glucose measurement system (Free Style®, DexCom® sensors, Enlite® sensors).
  Interventions: Other: CUTADIAB questionnaire

INTERVENTIONS:
Other: CUTADIAB questionnaire — During a regular diabetes follow-up consultation, the patient is asked to complete the CUTADIAB questionnaire on a tablet, entirely dedicated to the study

SUMMARY:
The use of technological tools in the treatment of diabetes has intensified and become common in recent years. Many of these systems adhere to the skin with an adhesive in place between 2 and 14 days. The objective of this study is to determine the prevalence and consequences of skin reactions to skin adhesive systems for the treatment of diabetes.

DETAILED DESCRIPTION:
The use of technological tools in the treatment of diabetes has intensified and become common in recent years. Many of these systems adhere to the skin with an adhesive in place for between 2 and 14 days, or even longer, depending on the system under consideration. Unfortunately, an increase in skin reactions has been observed in diabetic patients using these new technologies, sometimes leading to discontinuation. The number of studies evaluating the cutaneous tolerance of the patches used by these technologies is limited, so the prevalence of these skin intolerances is unknown.

The objective of this study is to determine the prevalence and consequences of skin reactions to skin adhesive systems for the treatment of diabetes. It will be implemented with the following design:

* observational, cross-sectional, multicentre study involving 4 Diabetology centres and over a period of 6 months.
* Establishment of an observatory on skin reactions to FreeStyle Libre® (FSL) and all other adhesive systems related to new technologies for the treatment of diabetes
* A questionnaire will be systematically proposed to the patients concerned, during the usual diabetes follow-up consultations made by all investigators.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* Adult (≥ 18 years old)
* All types diabetes (1, 2, other)
* Any patient who wears or has worn an adhesive system for the treatment of diabetes (insulin pump, and/or continuous glucose monitoring system) within the last 10 years.
* Seen consecutively in consultation
* Patient who was informed on the research and are not opposed to participation.

Exclusion Criteria:

* Illiteracy
* Refusal to participate in the study (refusals will be counted)
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major diabetic subjects, whatever the etiology of diabetes, using or having used in the last 10 years a system with skin adhesives, i.e. insulin patch pump (e.g. Omnipod®, cell Novo®), pump with externalized catheter (e.g. Minimed 640G®, Ypsopump®) or continuous glucose measurement system (Free Style®, Dexcom® sensors, Enlite® sensors).
Sampling Method: Non-Probability Sample
Enrollment: 851 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Percentage of skin intolerance to adhesives in diabetic patients | Single visit at day 0
  Percentage of skin intolerance in diabetic patients - all types of diabetes - using or having used in the last 10 years adhesive systems integrated into diabetes medical devices: patch insulin pump, pump with externalized catheter or continuous glucose measurement system.

SECONDARY OUTCOMES:
Prevalence of skin reactions by adhesive system | Single visit at day 0
  Skin intolerance in diabetic patients - all types of diabetes combined - using or having used adhesive systems integrated in diabetes medical devices, depending on the systems used
Consequences of skin reactions | Single visit at day 0
  Consequences of skin reactions (continuation / compliance / stopping / stopping then resuming and a delay time before resuming)
Percentage of positive responses to the question concerning patient approaches to avoid skin reaction | Single visit at day 0
  The patient is asked to answer the question "Do you use or have you used any tips to avoid or treat these skin manifestations" by choosing between the responses provided below (several possible items):
  * no
  * cortisone ointment on removal from the system
  * name of the ointment used:… ..
  * other ointment when removing the system
  * name of the ointment used:… ..
  * adhesive between skin and system
  * name of the adhesive used
  * other protection between the skin and the system (ointment, spray, etc.)
  * name of the protection used
  * stop using product before installation
  * change of the installation location of the system with the same reaction
  * change of the installation location of the system with improvement
  * stop using product before installation
Percentage of positive responses to the question concerning the delay of appearance of skin manifestation | Single visit at day 0
  The patient is asked to answer the question what time passed between the first use of the pump and the first appearance of skin manifestations by choosing between the responses provided below:
  * from the 1st installation
  * less than a week
  * less than a month
  * between 1 and 2 months
  * between 2 and 6 months
  * more than 6 months
Semiological description of skin lesions | Single visit at day 0
  The patient is asked to describe his skin manifestations by choosing between the responses provided below (several possible items):
  * redness
  * change in skin color (other than redness)
  * vesicles (blisters) / bubbles
  * peeling (loss of small pieces of skin)
  * it itches
  * it hurts
  * it flows
  * redness or bubbles are strictly localized under the adhesive
  * redness or bubbles overflow from the adhesive
  * infection (abscess or other) requiring treatment
  * antibiotic therapy / surgery (several items possible)
  * other (in full):
Evolution of lesions | Single visit at day 0
  The patient is asked to answer the question "How long is the reaction present?" by choosing between the responses provided below :
  * less than an hour
  * more than an hour and less than 24 hours
  * more than 24 hours and less than a week
  * more than a week and less than a month
  * more than a month
  * the reaction never went away

CONTACTS AND LOCATIONS:
Overall Officials: Agnès SOLA GAZAGNES, MD, Principal Investigator — AP-HP, Cochin Hospital, Department of Diabetology
Locations (4):
- France (4):
  - AP-HP, Lariboisière Hospital, Department of Diabetes and Endocrinology, Paris
  - AP-HP, Pitié-Salpêtrière Hospital, Diabetes and Metabolic Diseases Department, Paris
  - AP-HP, Cochin Hospital, Department of Diabetology, Paris
  - AP-HP, Bichat Hospital, Department of Diabetology, Endocrinology and Nutrition, Paris

REFERENCES:
- [Result] Diedisheim M, Pecquet C, Julla JB, Carlier A, Potier L, Hartemann A, Jacqueminet S, Vidal-Trecan T, Gautier JF, Dubois Laforgue D, Fagherazzi G, Roussel R, Larger E, Sola-Gazagnes A, Riveline JP. Prevalence and Description of the Skin Reactions Associated with Adhesives in Diabetes Technology Devices in an Adult Population: Results of the CUTADIAB Study. Diabetes Technol Ther. 2023 Apr;25(4):279-286. doi: 10.1089/dia.2022.0513. Epub 2023 Feb 24. PMID 36763338